CLINICAL TRIAL: NCT04914780
Title: The Effect of Training Performed Using Mobile Application on Care Requirements and Quality of Life in Women With Breast Cancer: Randomized Controlled Trial
Brief Title: The Effect of Training Given by Mobile Application to Women Undergoing Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayUHaticeTEZ
Record Dates: First submitted 2021-03-11; First posted 2021-06-07 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mobil Application; Quality of life; supportive Care Requirements
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 4 weeks training with mobile application
  Interventions: Behavioral: Education
- Control group (No Intervention): No intervention will be made for 4 weeks

INTERVENTIONS:
Behavioral: Education — Education intervention with mobile application for 4 weeks
  Arms: Intervention group

SUMMARY:
In a metanalysis study examining the effects of mobile health applications on the quality of life and psychological outcomes of patients with breast cancer, it was concluded that the quality of life increased, the level of self-efficacy was high, and the perceived stress, depression and anxiety were low compared to standard care. It has been stated that there is a need for well-designed randomized studies on the subject due to the heterogeneity of the study results. In a study examining the effects of exercise training given by mobile health application and traditional brochure on physical function, physical activity and quality of life in breast cancer patients, improvement was observed in both groups, but no significant difference was found between the groups. In the study conducted to evaluate the effect of the information transmitted via the mobile application on preoperative breast cancer patients, it was concluded that control patients who did not have access to additional information provided by the mobile application had significantly lower anxiety and depression scores at seven days before surgery compared to the intervention group, and thus, when less information was accessed. It has been reported that anxiety decreases. Surgical treatments applied to women with breast cancer, although there are different treatment options depending on the stage of the disease and the results of the diagnostic procedures; breast-conserving surgery (lumpectomy / tumorectomy, partial mastectomy, segmental mastectomy / quadranectomy) and non-breast-conserving surgery (simple mastectomy, bilateral mastectomy, skin-sparing mastectomy, nipple-sparing mastectomy, modified radical mastectomy, radical mastectomy). When the literature is examined; It was stated that negative emotions such as body image deterioration, decreased self-esteem, hopelessness, guilt, anxiety, and depression were experienced less in patients who underwent breast conserving surgery (BCS) compared to patients who received other breast surgical treatments. Compared to other patients, those who undergo BCS adapt better to the treatment and care process. There are some disadvantages for patients in BCS, which is preferred in the early stage, which aims to protect the integrity of the breast. Some of the disadvantages are the long-term treatment process, the expensive treatments and the difficult access for those living far from the radiotherapy treatment, which is mostly applied in large centers. In addition to these disadvantages, women experience intense psychosocial problems, symptoms experienced during the treatment process negatively affect their compliance with treatment and quality of life. In order to improve the affected quality of life, besides nursing interventions specially planned for each patient, trainings that will facilitate their adaptation to the disease during the diagnosis and treatment process should be planned.

DETAILED DESCRIPTION:
Breast cancer patients have many problems from different treatment processes and care needs to be met. Determining and supporting care needs affects the quality of life of patients. It is known that training provided by mobile applications enables patients with breast cancer to cope easily with their problems and increase their quality of life. Health needs to be individualized by shifting from institution- and physician-centered understanding to individual-centered healthcare service provision. There is no study in the literature evaluating the results of the training given specific to the supportive care needs with mobile application after surgery. The use of the mobile application that allows patient-centered supportive care for the education given to the patients reveals the difference of this study as it also includes interactive training. Mobile application to be created from educational content for patients with breast cancer; It aims to meet the holistic health care needs of women and to increase the quality of life by determining the individual care needs of women in the period after BCS. In this context, it is thought that the aim of reducing the care needs of patients and increasing the quality of life can be achieved with the education given to the patients. The mobile application includes maintaining and improving the health of women with breast cancer and offering solutions based on the literature for the problems they experience. It will be determined what the unmet needs of women with breast cancer that arise in different treatment processes, to what extent this process affects the quality of life of women and what solutions can be offered for these needs. In addition, the advantages and disadvantages of the mobile application method will be determined, and its effect on the patients' supportive care needs and quality of life will be revealed. The findings to be obtained, besides contributing to the literature, will reveal the educational needs of women with breast cancer and guide the treatment and care practices aimed at improving the quality of life. In addition, we aim to contribute to the development of mobile applications in the field of health by sharing our experiences with mobile application preparation. The mobile application developed after the study will be made available to all women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over,
* Breast Conserving Surgery is applied,
* Only diagnosed with breast cancer and not having metastases,
* Participating voluntarily in the research,
* Signed the informed consent form,
* Patients who have a smart phone on them or near them will be included in the study.

Exclusion Criteria:

* Not operated after the diagnosis of breast cancer and / or surgery other than Breast Conserving Surgery,
* Another type of cancer other than breast cancer,
* Having a disability to answer questions such as dementia, Alzheimer's, hearing and vision loss,
* Illiterate,
* Do not have a smart phone and / or do not know how to use it,
* Patients in the terminal period will not be included in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in supportive care needs at 4 weeks and 8 weeks | Baseline, 4 weeks and 8 weeks
  After the training given by the mobile application, the supportive care needs scores of the patients are checked.
  It has been stated that the DBGÖ-SF is a measurement tool with sufficient validity and reliability indicators. Your scale; There are 9 items in the "spiritual / psychological" sub-dimension and the minimum score from this dimension is 9; maximum score is 45. There are 10 items in the "Health system and information dimension" and the minimum score obtained from this dimension is 10; maximum score is 50. There are 5 items in the "Physical and daily life" dimension and the minimum score obtained from this dimension is 5; maximum score is 25. There are 4 items in the "patient care and support" dimension and the minimum score obtained from this dimension is 4; maximum score is 20. There are 3 items in the "sexuality" dimension and the minimum score obtained from this dimension is 3; maximum score is 15.

SECONDARY OUTCOMES:
Change from baseline in life quality at 4 weeks and 8 weeks | Baseline, 4 weeks and 8 weeks
  The quality of life scores of the patients are checked after the training given with the mobile application.
  Each area is calculated over a maximum of 20 points or 100 points. Which of these ratings will be used depends on the researcher. Calculations over 20 points are more commonly used in our country. The higher the score on the scale, the higher the quality of life. The correlation coefficients of the scale range between 0.49 and 0.78 (14th and 17th questions). When the Cronbach's alpha values are defined as values reflecting the homogeneity of the question scores with the field scores, the internal consistency of the sections and fields of WHOQOL-BREF (TR) was found to be quite high.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Medical Faculty Hospital Oncology Clinic, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the research is over